CLINICAL TRIAL: NCT03204968
Title: The Effect of Vagus Nerve Stimulation on the Inflammatory Response After Lung Lobectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otto Wagner Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Salama, MD, PhD, Otto Wagner Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Vagus Stimulation
Record Dates: First submitted 2017-06-23; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Inflammatory Response
Keywords: vagus nerve; Lung lobectomy
MeSH Terms: interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention)
- Treated (Active Comparator)
  Interventions: Device: Vagus nerve stimulation

INTERVENTIONS:
Device: Vagus nerve stimulation — transcutaneous Intermittent stimulation of the vagus nerve using neurostimulator V (Ducest®, Germany)
  Arms: Treated

SUMMARY:
Systemic inflammation is a potentially debilitating complication of thoracic surgeries that can result in significant physical and economic morbidity for afflicted patients. There is compelling evidence for the role of central nervous system in the regulation of systemic inflammatory responses through humoral mechanisms. Activation of afferent vagus nerve fibers by cytokines triggers anti-inflammatory responses. Direct electrical stimulation of the peripheral vagus nerve in vivo during lethal endotoxemia in rats inhibited Tumor necrosis factor (TNF) synthesis in liver preventing the development of shock. The vagal regulatory role of systemic inflammation after lung lobectomy is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Lung Lobectomy or pneumonectomy
* Adult
* Open surgery

Exclusion Criteria:

* Current infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2016-06-05 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
The postsurgical inflammatory response: the effect of vagus stimulation on proinflammatory interleukin concentrations | 3 time points: 24 hour prior to Operation (baseline), 1st and 4th postoperative day
  changes of serum Interleukin (IL-6, IL-10, IL-18, IL-1) concentrations in pg/ml from baseline and over the postsurgical course up to the 4th postoperative day in both study groups. The baseline is defined as the serum concentration of the target interleukins at 24 hours prior to surgery. Afterwards the changes in the interleukins concentrations will be measured on the 1st and 4th postoperative days in both groups in order to analyze the effect of vagus stimulation on the intensity of the postsurgical inflammatory response.

SECONDARY OUTCOMES:
The effect of vagus stimulation on changes in Serum C reactive protein (CRP) concentrations | 3 time points: 24 hour prior to Operation (baseline), 1st and 4th postoperative day
  changes of serum CRP concentrations in mg/L from baseline and over the postsurgical course up to the 4th postoperative day in both study groups. The baseline is defined as the serum concentration of CRP at 24 hours prior to surgery. Afterwards the changes in the interleukins concentrations will be measured on the 1st and 4th postoperative days in both groups in order to analyze the effect of vagus stimulation on the intensity of the postsurgical inflammatory response.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mueller, MD, PhD, Study Director — Otto Wagner Hospital; Mohamed Salama, MD, PhD, Principal Investigator — Otto Wagner Hospital
Locations (1):
- Department of Thoracic Surgery, Otto-Wagner Hospital, Vienna, Austria

REFERENCES:
- [Derived] Salama M, Akan A, Mueller MR. Transcutaneous Stimulation of Auricular Branch of the Vagus Nerve Attenuates the Acute Inflammatory Response After Lung Lobectomy. World J Surg. 2020 Sep;44(9):3167-3174. doi: 10.1007/s00268-020-05543-w. PMID 32358638
- See also: Related Info — https://www.researchgate.net/project/Postsurgical-Trauma-and-inflammatory-response